CLINICAL TRIAL: NCT01306487
Title: Correlation Between Visual Acuity and Recovery of Foveal Cone Microstructures After Macular Hole Surgery
Brief Title: Observation of Recovery of Foveal Cone Microstructures After Macular Hole Surgery
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Other Study IDs: Kyorineye002
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Macular Holes
Keywords: macular hole
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Macular hole patients: The patients who underwent vitreous surgery for idiopathic macular hole.
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Macular hole surgery
  Other Names: Optical coherence tomography

SUMMARY:
The objective is to determine whether a recovery of the microstructures of the foveal photoreceptors after macular hole (MH) closure is correlated with the best-corrected visual acuity (BCVA) is determined.

DETAILED DESCRIPTION:
Macular hole patients were evaluated by spectral domain optical coherence tomography (SD-OCT) to determine the integrity of the microstructures of the foveal photoreceptors. The inner segment/outer segment (IS/OS) junction, the external limiting membrane (ELM), and the cone outer segment tips (COST) line were determined preoperatively, and at 1, 3, 6, 9, and 12 months after the MH surgery. The correlation between the integrity of the foveal photoreceptor microstructures and the best-corrected visual acuity (BCVA) was determined.

ELIGIBILITY:
Inclusion Criteria:

* The patients had undergone surgery from March 2008 to August 2009 at Kyorin Eye Center
* Idiopathic macular hole patients with either a Stage 2, 3, or 4 according to the Gass classification

Exclusion Criteria:

* The presence of other retinal diseases including a treated rhegmatogenous retinal detachment, diabetic retinopathy
* High myopia with an axial length > 27.0 mm or refractive error > -8.0 diopters
* The patients followed for less than 6 months postoperatively

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with surgically-closed MHs after successful vitrectomy
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Foveal microstructure determined by optical coherence tomography | Preoperative and postoperative 1, 3, 6, 9, 12 months
  The integrity of the microstructures of the foveal photoreceptors; the inner segment/outer segment (IS/OS) junction, the external limiting membrane (ELM), and the cone outer segment tips (COST) line were determined by spectral domain optical coherence tomography.

SECONDARY OUTCOMES:
The visual acuity | Preoperative and postoperative 1, 3, 6, 9, 12 months
  Preoperative and postoperative best-corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan